CLINICAL TRIAL: NCT02868255
Title: Myeloid Derived Suppressor Cells Control by SIRP-alpha: Investigation in Hepatocellular Carcinoma
Brief Title: Myeloid Derived Suppressor Cells Control by Signal Regulatory Protein-alpha: Investigation in Hepatocellular Carcinoma
Acronym: MDScan
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC16_0156
Record Dates: First submitted 2016-06-16; First posted 2016-08-16 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Biobank analyses; Effect evaluation of the drug; patient-derived cells; SIRPα/CD47 expression
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and ascites will be analyzed for various cell populations by flow cytometry (different myeloid subsets including polymorphonuclear cells, MDSC and monocytes, T cell sub-populations including Tregs, CD8 and CD4 T cells, , B cells, and immature and mature NK cell). Myeloid infiltrate will be also evaluated by immunochemistry staining of CD68, CD163, CD206 and SIRPα of HCCs from the tumour bank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ascites: 30 inflammatory ascites of HCC patients (Collection of human samples ) Ascites will be selected only from HCC patients with an elevated protein level (ie inflammatory ascites) Puncture of ascites will be collected by paracentesis on HCC or ovarian cancer patients during their routine care These biological samples are affiliated with the biobank "hépato-gastroentérologie du CHU de Nantes" (declared under the reference DC-2011-1399).
  Interventions: Procedure: Collection of human samples
- Resections: 30 HCC resections (Collection of human samples ) Fragment of resected HCC will be obtained after surgery and histological analysis will be performed by the anatomo-pathology service These biological samples are affiliated with the biobank "hépato-gastroentérologie du CHU de Nantes" (declared under the reference DC-2011-1399).
  Interventions: Procedure: Collection of human samples
- blood samples: blood samples (Collection of human samples )will be collected prospectively for complementary functional analysis of peripheral These biological samples are affiliated with the biocollection "hépato-gastroentérologie du CHU de Nantes" (declared under the reference DC-2011-1399).
  Interventions: Procedure: Collection of human samples

INTERVENTIONS:
Procedure: Collection of human samples — Several types of samples will be used to test the effect of the drug candidate

SUMMARY:
project is to study and develop anti-Signal Regulatory Protein α (SIRPα) antibodies (Ab) as a new immunotherapy strategy in cancer.

Samples harvested from hepatocellular carcinoma (HCC) and ovarian cancer patients will be used in evaluation of the SIRP-CD47 expression and of the effect of the anti-human Signal Regulatory Protein (hSIRP) Ab on various cellular types from patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* adult
* HCC patients (all BCLC stages accepted)
* patient consent for the use of their biological samples

Exclusion Criteria:

* patient with other cancers
* hepatitis C or B positive
* HCC treatment by chemo-embolization under 3 months
* under Sorafenib treatment within the month prior to collection
* underage or under guardianship patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Several types of samples will be used to test the effect of the drug candidate: 30 inflammatory ascites of HCC patients, 30 HCC resections (both from CHU de Nantes), 30 HCC patient blood samples.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
evaluation of the SIRP/CD47 expression | baseline
  samples harvested from HCC and ovarian cancer patients will be used in evaluation of the SIRP-CD47 expression and of the effect of the anti-hSIRP Ab on various cellular types from patients

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ARCHAMBEAUD, Dr, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: No